CLINICAL TRIAL: NCT01063790
Title: The Effect of an Individualized Education Intervention Versus Usual Care on Pain Following Ambulatory Inguinal Hernia Repair
Brief Title: The Effect of an Individualized Education Intervention on Pain Following Inguinal Hernia Repair Surgery
Acronym: HREI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Mona Sawhney, PhD, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24390; 09-123c (Other: St. Michael's Hospital)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Pain
Keywords: Post-operative pain; inguinal hernia repair surgery; Patient education
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Pain Clinics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients undergoing elective inguinal hernia repair attend the pre-admission clinic no later than one week prior to surgery. During this visit they receive one-on-one pre-operative education from a registered nurse. It includes both verbal and written information. Verbal information provided to patients includes procedural information such as the admission process, and post-operative care in the post-anaesthetic care uni and day surgery unit. Post-discharge pain management information is minimal and consists of direction to not wait until the pain is severe before taking prescribed analgesics.
- Individualized Education (Experimental)
  Interventions: Behavioral: Individualized Education

INTERVENTIONS:
Behavioral: Individualized Education — The intervention consists of written information in the form of a booklet, an individualized face to face education session and two telephone support calls regarding post-discharge pain management, adverse effects of analgesics and common concerns about asking for help with pain.Participants in the intervention group will also receive two telephone support calls. The purpose of the telephone support calls is to readdress the information that patients received in the booklet and to clarify concerns regarding post-operative pain management that were discussed during the individualized education session.
  Other Names: inginal hernia repair; acute pain
  Arms: Individualized Education

SUMMARY:
Pain after inguinal hernia repair surgery is common with more than 50% of patients reporting moderate to severe acute pain following surgery. Analgesics are helpful in managing this pain but patients can be reluctant to take analgesics due to potential adverse effects such as nausea, vomiting or constipation. Patients may also be concerned about addiction to analgesics or they may believe that experiencing moderate to severe pain after surgery is to be expected.

The purpose of this study is to investigate the impact of an individualized education program regarding pain and management of adverse effects on pain after inguinal hernia repair surgery.

DETAILED DESCRIPTION:
There is clear evidence that patients who have undergone ambulatory inguinal hernia (IHR) repair have significant pain following surgery. Inguinal hernia repair has been identified as one of the most painful ambulatory surgery procedures, with 98% of patients reporting pain 24 hours following IHR surgery, and 54% of patients experiencing moderate to severe pain in the first 72 hours. Despite experiencing continued pain, patients do not always take the prescribed analgesics. Analgesics are helpful in managing post-operative pain but may have adverse effects, including nausea, vomiting or constipation, which are often not managed. Almost half of all patients who undergo ambulatory surgery experience these adverse effects with 45% experiencing constipation and 46% experiencing nausea and/or vomiting in the first 48 hours after surgery.

As well, patients may have concerns about addiction, or asking for help to manage their pain and may believe that moderate to severe pain is to be expected, contributes to healing and therefore is to be tolerated following surgery. Patients are expected to manage this pain and adverse effects of analgesics at home. Minimal research has been found regarding interventions to manage pain following ambulatory surgery, and none found specifically for patients undergoing inguinal hernia repair.

The purpose of this trial is to investigate the impact of an individualized pre-operative pain education intervention that includes a booklet with telephone support pre-operatively and after discharge home versus usual care for patients having IHR surgery. The primary outcome will be worst pain on movement in the past 24 hours and the secondary outcomes will be pain related interference, pain quality, analgesic use and adverse effects, and patient satisfaction and concerns with pain management.

ELIGIBILITY:
Inclusion Criteria:

* male
* able to speak, read and understand English,
* have telephone access.
* are scheduled for a unilateral inguinal hernia repair.

Exclusion Criteria:

* patients scheduled for a repeat IHR on the same surgical side
* patients who have emergency surgery.
* patients undergoing bilateral inguinal hernia repair.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is pain intensity using a 0 to 10 numeric rating scale. | Second post-operative day

SECONDARY OUTCOMES:
Secondary measures include: quality of pain, pain related interference, analgesic use, prevalence and intensity of adverse effects of analgesics, patient concerns regarding pain management, and adequacy of post-discharge information. | 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Judy Watt-Watson, RN, PhD, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada